CLINICAL TRIAL: NCT00657033
Title: A Randomized, Double Blind, Parallel Group, Multi-center Study to Investigate the Efficacy and Safety of Vardenafil Flexible Dose Versus Placebo in Males With Erectile Dysfunction, and Their Female Partners' Sexual Quality of Life.
Brief Title: Study to Investigate the Efficacy and Safety of Vardenafil Flexible Dose Versus Placebo in Males With Erectile Dysfunction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 100519
Record Dates: First submitted 2008-04-09; First posted 2008-04-14 (Estimated); Last update posted 2013-10-14 (Estimated); Status verified 2013-10

CONDITIONS: Erectile Dysfunction
Keywords: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Vardenafil Dihydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Levitra (Vardenafil, BAY38-9456)
- Arm 2 (Experimental)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levitra (Vardenafil, BAY38-9456) — BAY 38-9456 (Vardenafil) will be supplied as 5 mg tablets, 10 mg tablets, and 20 mg tablets.
  Arms: Arm 1
Drug: Placebo — Identical placebo tablets will be matched for each vardenafil dosage and will be indistinguishable from active treatment
  Arms: Arm 2

SUMMARY:
Study to investigate the efficacy and safety of vardenafil flexible dose versus placebo in males with erectile dysfunction, and their female partners' sexual quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Males who have had ED for at least six months according to the National Institutes of Health (NIH) Consensus Conference December 7-9, 1992 (inability to attain and/or maintain penile erection sufficient for satisfactory sexual performance).
* Stable, heterosexual relationship for more than 6 months.
* Males 18 years, and older.
* Written informed consent obtained.
* The subject and his female partner must make at least four attempts at sexual intercourse on four separate days during the untreated baseline period (according to the answer to the following question in the Patient Diary: "Was sexual activity initiated with the intention of intercourse?").
* At least 50% of attempts at sexual intercourse during the untreated baseline period must be unsuccessful, according to the following questions from the subject diary (at least one question should be answered "No"): "Were you able to achieve at least some erection (some enlargement of the penis)?"; "Were you able to insert your penis in your partner's vagina?"; "Did your erection last long enough for you to have successful intercourse?".

Exclusion Criteria:

A) Previous or current medical conditions:

* Any unstable medical, psychiatric, or substance abuse disorder that in the opinion of the Investigator is likely to affect the subject's ability to complete the study or precludes the subject's participation in the study.
* Presence of penile anatomical abnormalities (e.g. penile fibrosis or Peyronie's disease) which, in the Investigator's opinion, would significantly impair erectile function.
* Primary hypoactive sexual desire.
* Spinal cord injury.
* History of surgical prostatectomy (excluding TURP).
* Retinitis pigmentosa.
* Unstable angina pectoris.
* History of myocardial infarction, stroke or life-threatening arrhythmia within the prior 6 months.
* Uncontrolled atrial fibrillation/flutter at screening (ventricular response rate ≥ 100 bpm).
* Severe chronic or acute liver disease, history of moderate or severe hepatic impairment.
* Clinically significant chronic haematological disease which may lead to priapism such as sickle cell anemia and leukemia.
* Bleeding disorder.
* Significant active peptic ulcer disease.
* Resting hypotension (a resting systolic blood pressure of < 90 mm Hg) or hypertension (a resting systolic blood pressure > 170 mm Hg or a resting diastolic blood pressure > 110 mm Hg).
* History of malignancy within the past 5 years (other than squamous or basal cell skin cancer).
* NYHA Class III and IV heart failure.
* History of positive test for Hepatitis B surface antigen (HBsAg) or Hepatitis C.
* Symptomatic postural hypotension within 6 months of visit 1.

B) Concomitant medication:

* Subjects who are taking nitrates or nitric oxide donors.
* Subjects who take anticoagulants, except for antiplatelet agents.
* Subjects who are taking androgens.
* Subjects who are taking anti-androgens.
* Subjects who are taking the following inhibitors of cytochrome P450 3A4: very potent HIV protease inhibitors (ritonavir, indinavir), the anti-mycotic agents itraconazole and ketoconazole (topical forms are allowed) or erythromycin.
* Subjects who have received any investigational drug (including placebo) within 30 days of Visit 1.
* Use of any treatment for ED within 7 days of visit 1 or during the study, including oral medications, vacuum devices, constrictive devices, injections or urethral suppositories.
* Subjects who are taking alpha blockers

C) Abnormal laboratory values:

* Subjects who have a serum total testosterone level more than 25% below the age-adjusted lower limit of normal according to the range of the testing laboratory.
* Subjects with a serum creatinine > 3.0 mg/dl.
* Elevation of AST and/or ALT > 3 times the upper limit of normal.
* Diabetic subjects with an HbA1c>12%.

D) Other Exclusion Criteria:

* Subjects age 65 or older who in the judgment of the investigator can not be started on a 10 mg dose
* Subjects with a history of unresponsiveness to any PDE 5 Inhibitor treatment due to lack of efficacy or significant side effects leading to discontinuation of the PDE 5 Inhibitor treatment.
* Subjects unwilling to cease use of vacuum devices, intracavernosal injections, Viagra® or other therapy for ED during the study.
* Unwillingness of the subject or his partner to make 4 attempts at sexual intercourse on four separate days during the untreated baseline period.
* Subjects with known hypersensitivity to Vardenafil, Bay 38-9456 (also known as SB-782528) or any component of the investigational medication.
* Subjects who are illiterate or unable to understand the questionnaires or the Patient Diary.
* Partners who are illiterate or unable to understand the questionnaires.
* Subjects who are unwilling or unable to complete the Patient Diary.
* Subjects or partners who, in the opinion of the investigator, would be non-compliant with the visit schedule of study procedures.
* Subjects unwilling to refrain from consuming grapefruit juice or products containing grapefruit juice with study medication (Canada only).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2003-10; Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
The primary measures of efficacy in this study will be improved success of erection maintenance in men with ED and improvement in female partner's sexual quality of life. | Weeks 0 -12

SECONDARY OUTCOMES:
SEP3 at weeks 4 and 12 of treatment compared to placebo. | Weeks 4 and 12
Additional Patient Diary questions at 4 weeks, 8 weeks, 12 weeks, LOCF, and over entire treatment period compared to placebo. Per-subject success rates will be calculated as the number of successes divided by the number of sexual attempts with a resp | Weeks 4, 8 and 12
Global assessment question (GAQ) at weeks 4 and 12 of treatment compared to placebo | Weeks 4 and 12
Global confidence question (GCQ) at 12 weeks of treatment compared to placebo. | Week 12
The score for the IIEF questionnaire EF domain (IIEF-EF) at weeks 4, 12, and LOCF of treatment compared to placebo | Weeks 4 and 12
Scores from the Treatment Satisfaction Scale (TSS) -- Subject Active Medication module at week 12 and LOCF of treatment compared to placebo. The TSS is a self-report measure of subject and partner's satisfaction with various aspects of erectile function | Week 12
Scores from the mSLQQ-QOL at week 12 and LOCF of treatment compared to placebo | Week 12
Percentage of subjects achieving back to normal rates of erectile functioning (IIEF-EF > 25) at week 12 of treatment compared to placebo. | Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (25):
- United States (17):
  - Phoenix, Arizona
  - Beverly Hills, California
  - Irvine, California
  - Newport Beach, California
  - San Bernardino, California
  - San Diego, California
  - Trumbull, Connecticut
  - Jacksonville, Florida
  - Riverdale, Georgia
  - Greenbelt, Maryland
  - Lutherville, Maryland
  - Lawrenceville, New Jersey
  - New Brunswick, New Jersey
  - New York, New York
  - Charlotte, North Carolina
  - Statesville, North Carolina
  - Wilmington, North Carolina
- Canada (8):
  - Calgary, Alberta
  - Barrie, Ontario
  - Burlington, Ontario
  - Kitchener, Ontario
  - London, Ontario
  - Oakville, Ontario
  - Saskatoon, Saskatchewan
  - Victoria